CLINICAL TRIAL: NCT04649151
Title: A Phase 2/3, Randomized, Observer-Blind, Placebo-Controlled Study to Evaluate the Safety, Reactogenicity, and Effectiveness of mRNA-1273 SARS-CoV-2 Vaccine in Healthy Adolescents 12 to <18 Years of Age
Brief Title: A Study to Evaluate the Safety, Reactogenicity, and Effectiveness of mRNA-1273 Vaccine in Adolescents 12 to <18 Years Old to Prevent COVID-19
Acronym: TeenCove
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1273-P203; 2023-000382-14 (EudraCT Number)
Record Dates: First submitted 2020-11-30; First posted 2020-12-02 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; mRNA-1273.222 vaccine; SARS-CoV-2 VOC; SARS-CoV-2 VOC vaccine; Omicron; Variant; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1A is observer-blind. Participants will remain blinded until the initiation of Part 1B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- mRNA-1273 (Experimental): Part 1A (Blinded Phase): Participants will receive 2 intramuscular (IM) injections of mRNA-1273 (100 microgram [ug] each), 28 days apart, on Day 1 and Day 29.
  Part 1B (Open-Label Phase): Participants who cross over from placebo in Part 1A to Part 1B will receive 2 IM injections of mRNA-1273 (100 ug each), 28 days apart on Open Label Day 1 and Open Label Day 29.
  Part 2 (Open-Label): Participants will receive 2 IM injections of mRNA-1273 (50 ug each), 28 days apart, on Day 1 and Day 29 and may receive a booster dose on Day 149.
  Interventions: Biological: mRNA-1273
- Placebo (Placebo Comparator): Part 1A (Blinded Phase): Participants will receive 2 IM injections of mRNA-1273 matching placebo, 28 days apart, on Day 1 and Day 29.
  Interventions: Biological: Placebo
- mRNA-1273 BD (Experimental): Part 1C-1 (BD Phase): Participants will receive 1 IM injection of mRNA-1273 (50 ug) on BD-Day 1, 5 months after the last dose of Part 1A and 1B.
  Part 1C-2 (BD Phase): Participants will receive 1 IM injection of mRNA-1273 (50 ug) on BD-Day 1, at least 3 months post-last dose.
  Interventions: Biological: mRNA-1273
- mRNA-1273.222 (Experimental): Part 3 (Open-Label): Participants will receive up to 2 IM injections of mRNA-1273.222 (50 ug each), 6 months apart, on Day 1 and Day 181.
  Interventions: Biological: mRNA-1273.222

INTERVENTIONS:
Biological: mRNA-1273 — Sterile liquid for injection
  Arms: mRNA-1273; mRNA-1273 BD
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo
Biological: mRNA-1273.222 — Sterile solution for injection
  Arms: mRNA-1273.222

SUMMARY:
The mRNA-1273 vaccine is being developed to prevent COVID-19, the disease resulting from Severe Acute Respiratory Syndrome coronavirus (SARS-CoV-2) infection. The study is designed to primarily evaluate the safety, reactogenicity, and effectiveness of mRNA-1273 vaccine administered as primary series and a booster dose (BD) to an adolescent population. The study will also evaluate the safety and immunogenicity of an mRNA-1273.222 vaccine against the SARS-CoV- 2 omicron variant as a primary series.

DETAILED DESCRIPTION:
This is a Phase 2/3 study, with Part 1A (Blinded Phase), Part 1B (Open-label Observational Phase), Part 1C (Booster Dose [BD] Phase), which consists of Part 1C-1 and Part 1C-2, Part 2 (Open-Label), and Part 3 (Open-label). Participants in Part 1A are blinded to their treatment assignment, with participants receiving either 2 active mRNA-1273 vaccine doses or placebo. Part 1B of the study is designed to offer participants whose age group becomes Emergency Use Authorization (EUA) eligible to be unblinded so that participants who received placebo in Part 1A can request 2 doses of open-label mRNA-1273 vaccine. Part 1C-1 of the study will offer participants in Part 1A and Part 1B who are at least 5 months from the last dose, the option to request a homologous BD of mRNA-1273. Part 1C-2 is designed to provide a heterologous BD of mRNA-1273 to eligible participants who completed primary COVID-19 vaccination series with a non-Moderna vaccine under EUA and are at least 3 months from the last dose. Part 2 is an open-label design. Participants will receive 2 doses and may receive a booster dose of mRNA-1273 SARS-CoV-2 vaccine. Part 3 is an open-label design. Participants will receive up to 2 doses of mRNA-1273.222 vaccine.

Please access http://TeenCoveStudy.com for additional information, such as Study Overview, Participation, Site Locations along with contact numbers for each location for the study.

ELIGIBILITY:
Inclusion Criteria:

For Part 1A, Part 2 and Part 3:

* Participants 12 to <18 years of age at the time of consent (Screening Visit, Day 0) who, in the opinion of the Investigator, are in good general health based on review of medical history and screening physical examination.
* Investigator assessment that the participant, in the case of an emancipated minor, or parent(s)/legally acceptable representative(s) (LAR[s]) understand and is willing and physically able to comply with protocol-mandated follow up, including all procedures and provides written informed consent/assent.
* Body mass index (BMI) at or above the third percentile according to World Health Organization (WHO) Child Growth Standards at the Screening Visit (Day 0)
* Female participants of nonchildbearing potential may be enrolled in the study. Nonchildbearing potential is defined as premenarche or surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy).
* Female participants of childbearing potential may be enrolled in the study if the participant has a negative pregnancy test at Screening (Day 0), on the day of the first injection (Day 1), on the day of the second injection (Day 29 in Parts 1A and Part 2, and Day 181 in Part 3); has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first injection (Day 1); and has agreed to continue adequate contraception or abstinence through 3 months following the second injection (Day 29 in Part 1A and Part 2, and Day 181 in Part 3).

For Part 1B:

* Participants must have been previously enrolled in mRNA-1273-P203 study.
* Female participants of childbearing potential may be enrolled in the study if the participant has a negative pregnancy test on the day of the first injection (Open-Label-Day 1) and on the day of the second injection (Open-Label-Day 29).

For Part 1C-1 Homologous Booster Dose:

* Participants must have been previously enrolled in the mRNA-1273-P203 study, are actively participating in Part 1A or Part 1B and are least 5 months from the last dose.
* Female participants of childbearing potential may be enrolled in the study if the participant has a negative pregnancy test on the day of the first injection (BD-Day 1).

Part 1C-2 Heterologous Booster Dose:

* Male or female, 12 to < 18 years of age at the time of consent who, in the opinion of the investigator, is in good general health based on review of medical history and screening physical examination AND has completed non-Moderna primary COVID-19 vaccination series under EUA (for example, Pfizer) at least 3 months from consent.

Exclusion Criteria:

For Part 1A, Part 2, and Part 3:

* Has a known history of SARS-CoV-2 infection within 2 weeks prior to administration of investigational product (IP) or known close contact with anyone with laboratory-confirmed SARS-CoV-2 infection of COVID-19 within 2 weeks prior to administration of IP (Part 2 participants only). For Part 3 participants, known history of SARS-CoV-2 infection within 90 days prior to administration of IP or known close contact with anyone with laboratory-confirmed SARS-CoV-2 infection or COVID-19 within 90 days prior to administration of IP.
* Travel outside of the United States or home country (Part 2 and Part 3 only) in the 28 days prior to the Screening Visit (Day 0).
* Pregnant or breastfeeding
* Is acutely ill or febrile 24 hours prior to or at the Screening Visit (Day 0). Fever is defined as a body temperature ≥38.0°Celsius (C)/≥100.4°Farenheit (F). Participants who meet this criterion may have visits rescheduled within the relevant study visit windows. Afebrile participants with minor illnesses can be enrolled at the discretion of the Investigator.
* Prior administration of an investigational coronavirus (for example, SARS-CoV-2, SARS-CoV, Middle East Respiratory Syndrome [MERS-CoV]) vaccine
* Current treatment with investigational agents for prophylaxis against COVID-19
* Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation, or that could interfere with safety assessments or interpretation of results according to the Investigator's judgment
* Current use of any inhaled substance (for example, tobacco or cannabis smoke, nicotine vapors)
* History of chronic smoking (≥1 cigarette a day) within 1 year of the Screening Visit (Day 0)
* History of illegal substance use or alcohol abuse within the past 2 years. This exclusion does not apply to historical cannabis use that was formerly illegal in the participant's state but is legal at the time of screening.
* History of a diagnosis or condition that, in the judgment of the Investigator, may affect study endpoint assessment or compromise participant safety, specifically:

  * Congenital or acquired immunodeficiency, including human immunodeficiency virus (HIV) infection
  * Suspected active hepatitis
  * Has a bleeding disorder that is considered a contraindication to IM injection or phlebotomy
  * Dermatologic conditions that could affect local solicited AR assessments
  * History of anaphylaxis, urticaria, or other significant AR requiring medical intervention after receipt of a vaccine
  * Diagnosis of malignancy within the previous 10 years (excluding nonmelanoma skin cancer)
  * Febrile seizures
* Receipt of:

  * Any licensed vaccine within 28 days before the first dose of IP or plans for receipt of any licensed vaccine within 28 days before and/or after each dose of IP.
  * Systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to the day of enrollment (for corticosteroids, ≥20 mg/day prednisone equivalent). Topical tacrolimus is allowed if not used within 14 days prior to the day of enrollment. Participants may have visits rescheduled for enrollment if they no longer meet this criterion within the Screening Visit window. Inhaled, nasal, and topical steroids are allowed.
  * Intravenous blood products (red cells, platelets, immunoglobulins) within 3 months prior to enrollment
* Has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Screening Visit (Day 0) or plans to donate blood products during the study
* Participated in an interventional clinical study within 28 days prior to the Screening Visit (Day 0) or plans to do so while participating in this study
* Is an immediate family member or has a household contact who is an employee of the research center or otherwise involved with the conduct of the study

For Part 1C-1 and Part 1C-2:

* Pregnant or breastfeeding.
* Is acutely ill or febrile 24 hours prior to or at the Screening Visit (Day 0). Fever is defined as a body temperature ≥ 38.0°C/≥ 100.4°F. Participants who meet this criterion may have visits rescheduled within the relevant study visit windows. Afebrile participants with minor illnesses can be enrolled at the discretion of the investigator.
* Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation, or that could interfere with safety assessments or interpretation of results according to the investigator's judgment.
* History of a diagnosis or condition (after enrolment in Part 1A) that, in the judgment of the investigator, may affect study endpoint assessment or compromise participant safety:

  * Suspected active hepatitis
  * Has a bleeding disorder that is considered a contraindication to IM injection or phlebotomy
  * Dermatologic conditions that could affect local solicited AR assessments
  * History of anaphylaxis, urticaria, or other significant AR requiring medical intervention after receipt of a vaccine
  * Diagnosis of malignancy (excluding nonmelanoma skin cancer)
* Receipt of:

  • Any authorized or licensed vaccine within 28 days before the first dose of IP or plans for receipt of any licensed vaccine through 28 days following the last dose of IP or any seasonal influenza vaccine within 14 days before the first dose of IP or plans for receipt of any seasonal influenza vaccine 14 days following the last dose of IP.
* Participated in an interventional clinical study, other than mRNA-1273-P203 study, within 28 days prior to the Screening Visit (Day 0 [for Part 1C-1], BD-Day 0 [for Part 1C-2]) or plans to do so while participating in this study.

Part 1C-2 Heterologous Booster Dose:

* Has a known history of SARS-CoV-2 infection within 2 weeks prior to administration of IP or known close contact with anyone with laboratory-confirmed SARS-CoV-2 infection or COVID 19 within 2 weeks prior to administration of IP.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4328 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (52):
- United States (47):
  - Velocity Clinical Research - Banning, Banning, California
  - Paradigm Clinical Research, La Mesa, California
  - Altus Research - Hunt - PPDS, Lake Worth, Florida
  - Accel Research Sites - Nona Pediatric Center - ERN - PPDS, Orlando, Florida
  - Tekton Research - Georgia - PPDS, Chamblee, Georgia
  - IACT Health - Roswell - IACT - HyperCore - PPDS, Columbus, Georgia
  - Meridian Clinical Research - (Macon Georgia) - Platinum - PPDS, Macon, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Velocity Clinical Research - Boise - PPDS, Meridian, Idaho
  - Olivo Medical and Wellness Center, Chicago, Illinois
  - Velocity Clinical Research - Valparaiso, Valparaiso, Indiana
  - Meridian Clinical Research (Sioux City - Iowa), Sioux City, Iowa
  - Alliance for Multispecialty Research -El Dorado, El Dorado, Kansas
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Velocity Clinical Research - Metairie - PPDS, Metairie, Louisiana
  - University of Massachusetts Medical School, Molecu, Worcester, Massachusetts
  - Clinical Research Institute, Inc - CRN - PPDS, Minneapolis, Minnesota
  - Velocity Clinical Research - Gulfport - PPDS, Gulfport, Mississippi
  - Sundance Clinical Research - Platinum - PPDS, St Louis, Missouri
  - Meridian Clinical Research (Hastings-Nebraska) - Platinum - PPDS, Hastings, Nebraska
  - Quality Clinical Research - HyperCore - PPDS, Omaha, Nebraska
  - Meridian Clinical Research (Omaha-Nebraska) - Platinum - PPDS, Omaha, Nebraska
  - Velocity Clinical Research - Albuquerque - PPDS, Albuquerque, New Mexico
  - Child Healthcare Associates - East Syracuse, East Syracuse, New York
  - Meridian Clinical Research (Endwell-New York) - Platinum - PPDS, Endwell, New York
  - Velocity Clinical Research - Cincinnati - PPDS, Cincinnati, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute PC - CRN - PPDS, Tulsa, Oklahoma
  - Cyn3rgy Research - ClinEdge - PPDS, Gresham, Oregon
  - Velocity Clinical Research - Providence - PPDS, East Greenwich, Rhode Island
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Meridian Clinical Research - Charleston, SC, Charleston, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Benchmark Research, Austin, Texas
  - Coastal Bend Research Center, Corpus Christi, Texas
  - ACRC Trials, Frisco, Texas
  - DM Clinical Research - Kool Kids Pediatrics - ERN - PPDS, Houston, Texas
  - Clinical Trials of Texas, Inc. - PPDS, San Antonio, Texas
  - Tekton Research, San Antonio, Texas
  - Cope Family Medicine - Ogden Clinic - CCT, Bountiful, Utah
  - Wee Care Pediatrics - Kaysville, Kaysville, Utah
  - Cottonwood Pediatrics, Murray, Utah
  - South Ogden Family Medicine/Ogden Clinic - CCT Research, South Ogden, Utah
  - Alliance for Multispecialty Research, Syracuse, Utah
  - Advanced Clinical Research - Jordan Valley - ERN - PPDS, West Jordan, Utah
  - Meridian Clinical Research (Norfolk, Virginia), Norfolk, Virginia
  - Meridian Clinical Research - Family Practice Ports - Portsmouth - Platinum - PPDS, Portsmouth, Virginia
- Dominican Republic (5):
  - Caimed Dominicana S.A.S, Santo Domingo, Nacional
  - Hospital General Regional Dr. Marcelino Velez Santana, Santo Domingo, Nacional
  - Hospital Materno Infantil San Lorenzo de Los Mina, Santo Domingo, Nacional
  - Instituto Dermatologico y Cirugia de la Piel Dr. H Sede San Cristóbal, Santo Domingo, Nacional
  - Instituto Dominicano de Estudios Virologicos IDEV, Santo Domingo, Nacional

REFERENCES:
- [Derived] Figueroa AL, Torres D, Reyes-Acuna C, Matherne P, Yeakey A, Deng W, Xu W, Sigal Y, Chambers G, Olsen M, Girard B, Miller JM, Das R, Priddy F. Safety and immunogenicity of a single-dose omicron-containing COVID-19 vaccination in adolescents: an open-label, single-arm, phase 2/3 trial. Lancet Infect Dis. 2025 Feb;25(2):208-217. doi: 10.1016/S1473-3099(24)00501-2. Epub 2024 Sep 24. PMID 39332418
- [Derived] Ali K, Berman G, Zhou H, Deng W, Faughnan V, Coronado-Voges M, Ding B, Dooley J, Girard B, Hillebrand W, Pajon R, Miller JM, Leav B, McPhee R. Evaluation of mRNA-1273 SARS-CoV-2 Vaccine in Adolescents. N Engl J Med. 2021 Dec 9;385(24):2241-2251. doi: 10.1056/NEJMoa2109522. Epub 2021 Aug 11. PMID 34379915
- See also: Click here to access the website, http://TeenCoveStudy.com, for additional information for the study, such as Study Overview, Participation, Site Locations, along with contact numbers for each location for the study. — http://TeenCoveStudy.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included Part 1A as the Blinded Phase with participants remaining blinded until the initiation of Part 1B (open-label cross-over vaccination phase), and Parts 1C-1, 1C-2, 2, and 3 as open-label.
Pre-assignment Details: A per-protocol immunogenicity subset (PPIS) of randomly selected participants from study mRNA-1273-P301 (P301) (NCT04470427) aged 18-25 meeting pre-specified criteria (N=296) was used for comparison assessments of immune response.
  Study "Completed" and "Not Completed" data reported in the Participant Flow were collected from "Overall Study" (that is, as 1 period regardless if a booster dose was received).
Groups:
- Part 1A: mRNA-1273 100 μg: Participants received at least 1 of 2 doses of 100 micrograms (μg) mRNA-1273 by intramuscular (IM) injection (Day 1 and Day 29).
- Part 1A: Placebo: Participants received at least 1 of 2 doses of placebo matched to mRNA-1273 by IM injection (Day 1 and Day 29). Participants had the option to receive crossover vaccination with 100 μg mRNA-1273 in Part 1B.
- Part 1C-2: mRNA-1273 50 μg Booster Dose (BD): Participants who completed primary COVID-19 vaccination series with a non-Moderna vaccine under emergency use authorization (EUA), received a single BD of 50 μg mRNA-1273 IM injection on BD Day 1.
- Part 2: mRNA-1273 50 μg: Participants received at least 1 of 2 doses of 50 μg mRNA-1273 by IM injection (Day 1 and Day 29).
- Part 3: mRNA-1273.222 50 µg: Participants received 1 dose of mRNA-1273.222 50 µg by IM injection (Day 1). Some participants may have received a second dose of mRNA-1273.222 50 µg at approximately 6 months after the first dose (Day 181).
Period: Overall Study
Arm/Group | Part 1A: mRNA-1273 100 μg | Part 1A: Placebo | Part 1C-2: mRNA-1273 50 μg Booster Dose (BD) | Part 2: mRNA-1273 50 μg | Part 3: mRNA-1273.222 50 µg
Started | 2490 | 1243 | 155 | 52 | 388
Part 1: 1st Injection | 2486 | 1240 | 0 | 0 | 0
Part 1: 2nd Injection | 2480 | 1222 | 0 | 0 | 0
Part 2: 1st Injection | 0 | 0 | 0 | 52 | 0
Part 2: 2nd Injection | 0 | 0 | 0 | 50 | 0
Part 3: 1 Dose | 0 | 0 | 0 | 0 | 388
Part 3: 2 Doses | 0 | 0 | 0 | 0 | 335
Safety Analysis Set | 2486 | 1240 | 155 | 52 | 388
Solicited Safety Set | 2485 | 1240 | 125 | 52 | 387
PPIS | 340 | 0 | 136 | 46 | 373
Per Protocol (PP) Set for Efficacy | 2142 | 1044 | 0 | 0 | 0
Part 2 BD | 0 | 0 | 0 | 19 | 0
PPIS SARS-CoV-2 Positive (PPIS-Pos) | 0 | 0 | 0 | 44 | 372
Part 1C-1 BD | 1357 (Received vaccination with 100 μg mRNA-1273 in Part 1A prior to BD in Part 1C-1.) | 51 (Received crossover vaccination with 100 μg mRNA-1273 in Part 1B prior to BD in Part 1C-1.) | 0 | 0 | 0
Part 1B Crossover Vaccination | 0 | 96 (Received crossover vaccination with 100 μg mRNA-1273 in Part 1B after receiving placebo in Part 1A.) | 0 | 0 | 0
Part 1C-1 PPIS-Negative (Neg) | 267 | 0 | 0 | 0 | 0
Completed | 1274 | 74 | 143 | 41 | 358
Not Completed | 1216 | 1169 | 12 | 11 | 30
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 3
Not completed — Physician Decision | 10 | 0 | 0 | 1 | 1
Not completed — Protocol Deviation | 25 | 3 | 0 | 0 | 0
Not completed — Received another COVID-19 vaccine under EUA | 495 | 730 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 370 | 113 | 2 | 7 | 15
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 256 | 29 | 10 | 3 | 6
Not completed — Other than specified | 59 | 294 | 0 | 0 | 4
Not completed — Death | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Part 1A Randomization Set: All participants who were randomized. Parts 1C-2, 2, and 3 Safety Set: participants who received at least 1 dose of study drug in Study mRNA-1273-P203 (P203). Study mRNA-1273-P301 (P301) (NCT04470427) mRNA-1273 100 μg: PPIS of randomly selected participants from Study P301 aged 18-25 meeting pre-specified criteria.
Groups:
- Part 1A: mRNA-1273 100 μg: Participants were randomized to receive 2 doses of 100 μg mRNA-1273 by IM injection (Day 1 and Day 29).
- Part 1A: Placebo: Participants were randomized to receive 2 doses of placebo by IM injection (Day 1 and Day 29). Participants had the option to receive crossover vaccination with 100 μg mRNA-1273 in Part 1B.
- Part 1C-2: mRNA-1273 50 μg BD: Participants who completed primary COVID-19 vaccination series with a non-Moderna vaccine under EUA, received a single booster of 50 μg mRNA-1273 IM injection on BD Day 1.
- Part 3: mRNA-1273.222 50 µg: Participants received 1 dose of mRNA-1273.222 50 µg by IM injection (Day 1). Participants may have received a second dose of mRNA-1273.222 50 µg at approximately month 6 after the first dose (Day 181).
- Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg: Participants (young adults; 18-25 years of age) received 100 μg mRNA-1273 on a 2 injection schedule in Study mRNA-1273-P301 (P301).
- Total: Total of all reporting groups
Arm/Group | Part 1A: mRNA-1273 100 μg | Part 1A: Placebo | Part 1C-2: mRNA-1273 50 μg BD | Part 2: mRNA-1273 50 μg | Part 3: mRNA-1273.222 50 µg | Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg | Total
Number analyzed (Participants) | 2490 | 1243 | 155 | 52 | 388 | 296 | 4624
Age, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics data of participants enrolled in Study mRNA-1273-P301 have been reported separately.
  Participants
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P203: number analyzed (Participants) | 2490 | 1243 | 155 | 52 | 388 | 0 | 4328
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P203: Adolescents (12-17 years) | 2490 | 1243 | 155 | 52 | 388 | 0 | 4328
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P203: Adults (18-64 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P301: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 296 | 296
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P301: Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P301: Adults (18-64 years) | 0 | 0 | 0 | 0 | 0 | 296 | 296
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics data of participants enrolled in Study mRNA-1273-P301 have been reported separately.
  Participants
    Sex Data for Participants Enrolled in Study mRNA-1273-P203: number analyzed (Participants) | 2490 | 1243 | 155 | 52 | 388 | 0 | 4328
    Sex Data for Participants Enrolled in Study mRNA-1273-P203: Female | 1206 | 607 | 78 | 26 | 185 | 0 | 2102
    Sex Data for Participants Enrolled in Study mRNA-1273-P203: Male | 1284 | 636 | 77 | 26 | 203 | 0 | 2226
    Sex Data for Participants Enrolled in Study mRNA-1273-P301: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 296 | 296
    Sex Data for Participants Enrolled in Study mRNA-1273-P301: Female | 0 | 0 | 0 | 0 | 0 | 153 | 153
    Sex Data for Participants Enrolled in Study mRNA-1273-P301: Male | 0 | 0 | 0 | 0 | 0 | 143 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics data of participants enrolled in Study mRNA-1273-P301 have been reported separately.
  Participants
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P203: number analyzed (Participants) | 2490 | 1243 | 155 | 52 | 388 | 0 | 4328
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P203: Hispanic or Latino | 280 | 152 | 37 | 14 | 367 | 0 | 850
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P203: Not Hispanic or Latino | 2190 | 1079 | 116 | 36 | 21 | 0 | 3442
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P203: Unknown or Not Reported | 20 | 12 | 2 | 2 | 0 | 0 | 36
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P301: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 296 | 296
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P301: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 78 | 78
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P301: Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 216 | 216
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P301: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics data of participants enrolled in Study mRNA-1273-P301 have been reported separately.
  Participants
    Race Data for Participants Enrolled in Study mRNA-1273-P203: number analyzed (Participants) | 2490 | 1243 | 155 | 52 | 388 | 0 | 4328
    Race Data for Participants Enrolled in Study mRNA-1273-P203: White | 2087 | 1043 | 115 | 30 | 39 | 0 | 3314
    Race Data for Participants Enrolled in Study mRNA-1273-P203: Black or African American | 83 | 42 | 23 | 18 | 126 | 0 | 292
    Race Data for Participants Enrolled in Study mRNA-1273-P203: Asian | 143 | 80 | 3 | 3 | 0 | 0 | 229
    Race Data for Participants Enrolled in Study mRNA-1273-P203: American Indian or Alaska Native | 12 | 7 | 1 | 0 | 1 | 0 | 21
    Race Data for Participants Enrolled in Study mRNA-1273-P203: Native Hawaiian or Other Pacific Islander | 3 | 0 | 0 | 0 | 0 | 0 | 3
    Race Data for Participants Enrolled in Study mRNA-1273-P203: Multiple | 118 | 50 | 9 | 0 | 3 | 0 | 180
    Race Data for Participants Enrolled in Study mRNA-1273-P203: Other | 27 | 9 | 4 | 0 | 219 | 0 | 259
    Race Data for Participants Enrolled in Study mRNA-1273-P203: Not Reported | 11 | 11 | 0 | 0 | 0 | 0 | 22
    Race Data for Participants Enrolled in Study mRNA-1273-P203: Unknown | 6 | 1 | 0 | 1 | 0 | 0 | 8
    Race Data for Participants Enrolled in Study mRNA-1273-P301: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 296 | 296
    Race Data for Participants Enrolled in Study mRNA-1273-P301: White | 0 | 0 | 0 | 0 | 0 | 207 | 207
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Black or African American | 0 | 0 | 0 | 0 | 0 | 29 | 29
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Asian | 0 | 0 | 0 | 0 | 0 | 30 | 30
    Race Data for Participants Enrolled in Study mRNA-1273-P301: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 2 | 2
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Multiple | 0 | 0 | 0 | 0 | 0 | 14 | 14
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Other | 0 | 0 | 0 | 0 | 0 | 8 | 8
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Not Reported | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs)
Description: Solicited ARs (local and systemic) were collected in an electronic diary (eDiary). Local ARs included injection site pain, injection site erythema (redness), injection site swelling/induration (hardness), and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs included fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. Solicited ARs considered causally related to injection were graded 1-4 (per Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials); lower score indicated lower severity, and higher score indicated greater severity. Investigator reviewed if the solicited AR was recorded as an adverse event (AE) as detailed in the AE section. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the AE section.
Time Frame: 7 days post-vaccination
Population: Solicited Safety Set included participants who received at least 1 dose of study drug and contributed any solicited AR data.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1A: mRNA-1273 100 μg: Participants received at least 1 of 2 doses of 100 μg mRNA-1273 by IM injection (Day 1 and Day 29).
- Part 1A: Placebo: Participants received at least 1 of 2 doses of placebo matched to mRNA-1273 100 μg by IM injection (Day 1 and Day 29).
- Part 1C-1: mRNA-1273 50 µg BD: Participants received mRNA-1273 100 µg in blinded or cross-over phase (Parts 1A or 1B) and then a single BD of 50 μg mRNA-1273 IM injection on BD Day 1 in Part 1 C-1.
- Part 1C-2: mRNA-1273 50 μg BD: Participants who completed primary COVID-19 vaccination series with a non-Moderna vaccine under EUA, received a single BD of 50 μg mRNA-1273 IM injection on BD Day 1.
- Part 2: mRNA-1273 50 μg First Injection: Participants received 1 dose of 50 μg mRNA-1273 by IM injection (Day 1).
- Part 2: mRNA-1273 50 μg Second Injection: Participants received 2nd dose of 50 μg mRNA-1273 by IM injection (Day 29).
- Part 2: mRNA-1273 50 μg BD: Participants received open-label mRNA-1273 50 μg in Part 2 and then a single BD of 50 μg mRNA-1273 IM injection on BD Day 1 in Part 2.
- Part 3: mRNA-1273.222 50 μg 1 Dose: Participants received 1 dose of mRNA-1273.222 50 μg by IM injection (Day 1).
Arm/Group | Part 1A: mRNA-1273 100 μg | Part 1A: Placebo | Part 1C-1: mRNA-1273 50 µg BD | Part 1C-2: mRNA-1273 50 μg BD | Part 2: mRNA-1273 50 μg First Injection | Part 2: mRNA-1273 50 μg Second Injection | Part 2: mRNA-1273 50 μg BD | Part 3: mRNA-1273.222 50 μg 1 Dose
Number analyzed (Participants) | 2485 | 1240 | 1351 | 125 | 52 | 46 | 19 | 387
Participants
  Grade 1 | 586 | 585 | 627 | 42 | 25 | 18 | 7 | 145
  Grade 2 | 1250 | 293 | 501 | 48 | 16 | 9 | 0 | 62
  Grade 3 | 627 | 59 | 150 | 9 | 1 | 3 | 1 | 25
  Grade 4 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Any Solicited (Grade 1-4) | 2466 | 938 | 1278 | 99 | 42 | 30 | 8 | 233

2. Primary Outcome: Number of Participants With Unsolicited AEs
Description: An unsolicited AE was any AE reported by the participant that was not specified as a solicited AR in the protocol or was specified as a solicited AR but started outside the protocol-defined period for reporting solicited ARs (onset after Day 7 of dosing). An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result or other safety assessment, including one that worsened from baseline and was considered clinically significant by the Investigator was recorded as an AE.
  Non-serious SARs persisting beyond 7 days, leading to discontinuation, or medically attended were classified as AEs in Part 1/2 but not in Part 3. COVID-19/SARS-CoV-2 infections were AEs in Part1/2 but were considered clinical events for efficacy in Part 3 and not AEs.
  A Summary of SAEs and nonserious AEs ("Other"), regardless of causality, is located in the AE section.
Time Frame: Up to 28 days post-vaccination
Population: Safety Set: participants who received at least 1 dose of study drug. As prespecified in the protocol, Part 1B was not assessed for this outcome measure. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: mRNA-1273 100 μg | Part 1A: Placebo | Part 1C-1: mRNA-1273 50 µg BD | Part 1C-2: mRNA-1273 50 μg BD | Part 2: mRNA-1273 50 μg | Part 2: mRNA-1273 50 μg BD | Part 3: mRNA-1273.222 50 μg 1 Dose
Number analyzed (Participants) | 2486 | 1240 | 1405 | 155 | 52 | 19 | 388
Participants | 582 | 237 | 209 | 19 | 10 | 2 | 52

3. Primary Outcome: Part 1A Geometric Mean Value of Serum Pseudovirus Neutralizing Antibody (nAb) ID50 Titers From Study P203 Vaccine Recipients at Day 57 Compared With Those From Young Adult (18 to 25 Years of Age) Vaccine Recipients (Day 57) in Study P301
Description: Pseudovirus nAb ID50 titers were measured using pseudovirus neutralization assay (PsVNA) assay. Antibody values reported as below the lower limit of quantification (LLOQ) were replaced by 0.5*LLOQ. Values greater than the upper limit of quantification (ULOQ) were replaced by the ULOQ if actual values were not available (LLOQ: 18.5 arbitrary units (AU)/milliliter (mL), ULOQ: 45118 AU/mL). Antibody levels were analyzed using an analysis of covariance (ANCOVA) model with the group variable (adolescents in P203 and young adults in P301) as fixed effect. PPIS P301: randomly selected participants from Study P301 aged 18-25 meeting pre-specified criteria were used for comparison assessments of immune response.
Time Frame: Day 57 Study P203/Day 57 Study P301
Population: Part 1A PPIS: randomized participants who were selected for the Immunogenicity Subset, received planned doses of study drug per schedule, complied with immunogenicity testing schedule, and had no major protocol deviations that impacted key or critical data. Participants who were seropositive at baseline were excluded from the PPIS. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg: Participants (young adults; 18-25 years of age) received 100 μg mRNA-1273 on a 2 injection schedule in Study mRNA-1273-P301 (P301).
Arm/Group | Part 1A: mRNA-1273 100 μg | Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg
Number analyzed (Participants) | 340 | 295
titer | 1401.670 [1276.218 to 1539.453] | 1299.855 [1175.380 to 1437.511]
Statistical Analysis 1: Comparison: Part 1A: mRNA-1273 100 μg vs Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg; Test type: Non-Inferiority — The noninferiority of Geometric Mean value (based on geometric least squares means [GLSM]) was considered demonstrated if: The lower bound of the 95% confidence interval (CI) of the geometric mean ratio (GMR) was >0.667 based on the noninferiority margin of 1.5, and the GMR point estimate ≥0.8 (minimum threshold); GMR = 1.078, 95% CI 2-sided [0.940 to 1.237] — GMR of P203 vs P301

4. Primary Outcome: Part 1A Seroresponse Rate (SRR) for Serum Pseudovirus nAb ID50 in Study P203 Vaccine Recipients at Day 57 Compared With Those From Young Adult (18 to 25 Years of Age) Vaccine Recipients (Day 57) in Study P301
Description: Percentage of participants with seroresponse for pseudovirus nAb ID50 measured using PsVNA assay are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4*LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ (LLOQ: 18.5 AU/mL), ULOQ: 45118 AU/mL).
  PPIS P301: randomly selected participants from Study P301 aged 18-25 meeting pre-specified criteria were used for comparison assessments of immune response.
Time Frame: Day 57 Study P203/Day 57 Study P301
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1A: mRNA-1273 100 μg | Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg
Number analyzed (Participants) | 340 | 295
percentage of participants | 98.8 [97.0 to 99.7] | 99.0 [97.1 to 99.8]
Statistical Analysis 1: Comparison: Part 1A: mRNA-1273 100 μg vs Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg; Test type: Non-Inferiority — Noninferiority margin of 10%. Lower bound of the 95% CI of the SRR difference >-10%. and a point estimator >-5% (minimum threshold); percentage difference = -0.2, 95% CI 2-sided [-2.1 to 1.9] — SRR difference of P203 vs P301

5. Primary Outcome: Part 1C-1 Geometric Mean Concentration (GMC) of Serum Pseudovirus nAb Against the Original Strain After the BD in Study P203 at BD Day 29 Compared With Those From Young Adult (18 to 25 Years of Age) Vaccine Recipients (Day 57) in Study P301
Description: Pseudovirus nAb were measured using PsVNA assay. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available (LLOQ: 10, ULOQ: 281600). PPIS P301: randomly selected participants from study P301 aged 18-25 meeting pre-specified criteria and SARS-CoV-2 negative were used for comparison assessments of immune response.
Time Frame: BD Day 29 Study P203/Day 57 Study P301
Population: Part 1C-1 PPIS-Neg: participants were baseline (pre-dose 1 of part 1A) SARS-CoV-2 negative, had BD-Day 1 and BD-Day 29 Ab assessment, had no major protocol deviations, did not receive off-study COVID-19 vaccination prior to BD-Day 29 visit, received 2 doses of mRNA-1273 in the Blinded Phase per schedule, received BD, and were pre-booster SARS-CoV2 negative. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: arbitrary units (AU)/mL
Groups:
- Part 1C-1: mRNA-1273 50 µg BD: Participants received mRNA-1273 100 µg in blinded or cross-over phase (Parts 1A or 1B) and then a single BD of 50 μg mRNA-1273 IM injection on BD Day 1 in Part 1C-1.
Arm/Group | Part 1C-1: mRNA-1273 50 µg BD | Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg
Number analyzed (Participants) | 264 | 294
arbitrary units (AU)/mL | 7102.0 [6553.2 to 7696.8] | 1400.4 [1272.7 to 1541.0]
Statistical Analysis 1: Comparison: Part 1C-1: mRNA-1273 50 µg BD vs Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg; Test type: Non-Inferiority — The lower bound of the 95% CI of noninferiority margin of 1.5. GMR point estimate >=0.8 (minimum threshold); GMR = 5.071, 95% CI 2-sided [4.477 to 5.745] — GMR of GMC at BD-Day 29 P203 vs GMC at Day 57 P301

6. Primary Outcome: Part 1C-1 SRR of Serum Pseudovirus nAb Against the Original Strain After the BD in Study P203 at BD Day 29 Compared With Those From Young Adult (18 to 25 Years of Age) Vaccine Recipients (Day 57) in Study P301
Description: Percentage of participants with seroresponse for pseudovirus nAb measured using PsVNA assay are reported. Seroresponse relative to pre-Dose 1 (baseline) at a participant level was defined as a change from below the LLOQ to equal or above 4 * LLOQ, or at least a 4-fold-rise if baseline was equal to or above LLOQ (LLOQ: 10 AU/mL, ULOQ: 281600 AU/mL). PPIS P301: randomly selected participants from Study P301 aged 18-25 meeting pre-specified criteria and SARS-CoV-2 negative were used for comparison assessments of immune response.
Time Frame: BD Day 29 Study P203/Day 57 Study P301
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1C-1: mRNA-1273 50 µg BD | Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg
Number analyzed (Participants) | 264 | 294
percentage of participants | 100.0 [98.6 to 100.0] | 99.3 [97.6 to 99.9]
Statistical Analysis 1: Comparison: Part 1C-1: mRNA-1273 50 µg BD vs Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg; Test type: Non-Inferiority — Noninferiority margin of 10%. Lower bound of the 95% CI of the SRR difference >-10%; SRR Difference = 0.7, 95% CI 2-sided [-0.8 to 2.4] — SRR difference of P203 BD-Day 29 vs P301 Day 57

7. Primary Outcome: Part 3 GMC of nAb Post Dose 1 mRNA 1273.222 Against Omicron BA.4/BA.5 Compared With Those From Young Adult (18 to 25 Years of Age) Vaccine Recipients (Day 57) in Study P301
Description: Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available (LLOQ: 103 AU/mL, ULOQ: 28571 AU/mL). ANCOVA model with the group variable (adolescents in P203 and young adults in P301) as fixed effect. PPIS P301: randomly selected participants from Study P301 aged 18-25 meeting pre-specified criteria and SARS-CoV-2 negative were used for comparison of immune response.
Time Frame: Day 29 Study P203/Day 57 Study P301
Population: Part 3 PPIS-Pos: participants received Dose 1 of mRNA-1273.222, had Day 29 antibody assessments, no major protocol deviations, did not receive off-study COVID-19 vaccination prior to Day 29, SARS-CoV-2 positive at Baseline. 'Overall number of participants analyzed' = participants evaluable for the endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 3: mRNA-1273.222 50 µg | Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg
Number analyzed (Participants) | 372 | 294
AU/mL | 2727.8 [2558.7 to 2908.1] | 56.6 [52.7 to 60.8]
Statistical Analysis 1: Comparison: Part 3: mRNA-1273.222 50 µg vs Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg; Test type: Superiority — The superiority of GMC (based on GLSM] was considered demonstrated if: The lower bound of the 95% CI of the GMR was >1; GMR = 48.191, 95% CI 2-sided [43.765 to 53.065] — GMR of P203 vs P301

8. Primary Outcome: Part 1C-2 GMC of Post-booster Pseudovirus nAb Against Ancestral Strain at BD Day 29
Description: Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available (LLOQ: 10 AU/mL, ULOQ: 111433 AU/mL).
Time Frame: BD Day 29
Population: Part 1C-2 PPIS: all randomized participants who received BD in Part 1C-2, had BD-Day 29 Ab assessment, had no major protocol deviations that impacted key or critical data, and did not receive off-study COVID-19 vaccination prior to BD-Day 29 visit. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1C-2: mRNA-1273 50 μg BD
Number analyzed (Participants) | 134
AU/mL | 9433.4 (8496.8) [8496.8 to 10473.3]

9. Primary Outcome: Part 2 GMC of the Pseudovirus nAb Against Ancestral Strain at Day 57
Description: as for outcome 8
Time Frame: Day 57
Population: Part 2 PPIS: all randomized participants who received at least 1 dose of the planned study drug, had Ab assessment for the analysis endpoint, and had no major protocol deviations that could impact key or critical data.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 2: mRNA-1273 50 μg
Number analyzed (Participants) | 46
AU/mL | 7351.5 (5621.7) [5621.7 to 9613.7]

10. Primary Outcome: Part 3 GMC of nAb Post Dose 1 mRNA 1273.222 Against SARS-CoV-2 Ancestral Strain Compared With Those From Young Adult (18 to 25 Years of Age) Vaccine Recipients (Day 57) in Study P301
Description: Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available (LLOQ: 10 AU/mL, ULOQ: 111433 AU/mL). ANCOVA model with the group variable (adolescents in P203 and young adults in P301) as fixed effect. PPIS P301: randomly selected participants from Study P301 aged 18-25 meeting pre-specified criteria and SARS-CoV-2 negative were used for comparison of immune response.
Time Frame: Day 29 Study P203/Day 57 Study P301
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 3: mRNA-1273.222 50 µg | Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg
Number analyzed (Participants) | 371 | 295
AU/mL | 7603.9 [7004.6 to 8254.6] | 1692.3 [1543.4 to 1855.5]
Statistical Analysis 1: Comparison: Part 3: mRNA-1273.222 50 µg vs Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg; Test type: Non-Inferiority — The noninferiority of Geometric Mean value (based on GLSM) was considered demonstrated if: The lower bound of the 95% CI of the GMR was >0.667 based on the noninferiority margin of 1.5, and the GMR point estimate ≥0.8 (minimum threshold); GMR = 4.493, 95% CI 2-sided [3.972 to 5.083] — GMR of GMC at BD-Day 29 P203 vs GMC at Day 57 P301

11. Primary Outcome: Part 2 SRR of Pseudovirus nAb Against Ancestral Strain
Description: Percentage of participants with seroresponse for pseudovirus nAb measured using PsVNA assay are reported. Seroresponse relative to pre-Dose 1 (baseline) at a participant level was defined as a change from below the LLOQ to equal or above 4 * LLOQ, or at least a 4-fold-rise if baseline was equal to or above the LLOQ (LLOQ: 10 AU/mL, ULOQ: 111433 AU/mL).
Time Frame: Day 57
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: mRNA-1273 50 μg
Number analyzed (Participants) | 46
percentage of participants | 91.3 (79.2) [79.2 to 97.6]

12. Primary Outcome: Number of Participants With SAEs, AEs of Special Interest (AESIs), Medically Attended AEs (MAAEs), and AEs Leading to Study Discontinuation
Description: SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AESIs were identified based upon medical concepts that may be related to COVID-19 or were of interest in COVID-19 vaccine safety surveillance. MAAE was an AE that led to an unscheduled visit to a healthcare practitioner, included visits to a study site for unscheduled assessments (for example, abnormal laboratory follow-up, and visits to healthcare practitioners external to the study site [for example, urgent care, primary care physician]). Non-serious SARs persisting beyond 7 days, leading to discontinuation, or medically attended were defined as AEs in Part 1/2 but not in Part 3. COVID-19/SARS-CoV-2 infections were AEs in Part 1/2 but were considered clinical events for efficacy in Part 3 and not AEs.
Time Frame: Day 1 up to Day 751
Population: Participants who received at least 1 dose of mRNA-1273 were included in the analysis. 'Overall number of participants analyzed' = participants evaluable for this endpoint. Note: Part 3 is presented for overall study for this assessment (AE section presents AEs separately for 1 dose and second dose).
Measure: Count of Participants; unit: Participants
Groups:
- Part 1B: mRNA-1273 100 μg: Participants previously received 2 doses of placebo in the blinded phase and then received crossover vaccination with 100 μg of mRNA-1273.
- Part 3: mRNA-1273.222 50 μg: Participants received 1 dose of mRNA-1273.222 50 μg by IM injection (Day 1). Some participants may have received a second dose of mRNA-1273.222 50 μg at approximately 6 months after the first dose (Day 181).
Arm/Group | Part 1A: mRNA-1273 100 μg | Part 1B: mRNA-1273 100 μg | Part 1C-1: mRNA-1273 50 µg BD | Part 1C-2: mRNA-1273 50 μg BD | Part 2: mRNA-1273 50 μg | Part 2: mRNA-1273 50 μg BD | Part 3: mRNA-1273.222 50 μg
Number analyzed (Participants) | 2486 | 96 | 1408 | 155 | 52 | 19 | 388
Participants
  SAEs | 21 | 2 | 9 | 3 | 0 | 0 | 16
  AESIs | 17 | 0 | 9 | 1 | 0 | 0 | 3
  MAAEs | 1040 | 31 | 541 | 45 | 12 | 7 | 183
  AEs Leading to Study Discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 1

13. Secondary Outcome: Part 1A Number of Participants With a SARS-CoV-2 Infection (Symptomatic or Asymptomatic)
Description: SARS-CoV-2 infection was defined in participants with negative SARS-CoV-2 status at baseline: bAb level against SARS-CoV-2 nucleocapsid protein negative at Day 1, that became positive postbaseline; or positive postbaseline.
Time Frame: Day 43 (14 days after second injection) up to a median follow up of 2.5 months after second injection
Population: Part 1A PP Set for Efficacy: all randomized participants who received planned doses of study drug, had no immunologic or virologic evidence of prior COVID-19, and had no major protocol deviations that impact key or critical efficacy data.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: mRNA-1273 100 μg | Part 1A: Placebo
Number analyzed (Participants) | 2142 | 1044
Participants | 22 | 25
Statistical Analysis 1: Comparison: Part 1A: mRNA-1273 100 μg vs Part 1A: Placebo; Test type: Other — The 95% CI of the ratio was calculated using the exact method conditional upon the total number of cases, adjusting for person-years; VE; Vaccine efficacy (VE, percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo); VE = 60.3, 95% CI 2-sided [26.6 to 78.6]

14. Secondary Outcome: Part 1A Number of Participants With Asymptomatic SARS-CoV-2 Infection
Description: Asymptomatic SARS-CoV-2 infection was defined as absence of symptoms and a positive RT-PCR or serology test (bAb levels against SARS-CoV-2 nucleocapsid protein) post dosing in participants who did not have an infection at baseline or pre-Dose 1.
Time Frame: Day 43 (14 days after second injection) up to a median follow up of 2.5 months after second injection
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: mRNA-1273 100 μg | Part 1A: Placebo
Number analyzed (Participants) | 2142 | 1044
Participants | 20 | 16
Statistical Analysis 1: Comparison: Part 1A: mRNA-1273 100 μg vs Part 1A: Placebo; Test type: Other — [test comment as in outcome 13, analysis 1]; VE; VE (percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo); VE = 43.5, 95% CI 2-sided [-16.5 to 72.2]

15. Secondary Outcome: Part 1A Number of Participants With a First Occurrence of Symptomatic COVID-19
Description: COVID-19 was defined as symptomatic disease based on the following criteria: participants experienced at least 2 of the following systemic symptoms: fever (≥ 38ºC/≥ 100.4ºF), chills, myalgia, headache, sore throat, new olfactory and taste disorder(s); or experienced at least 1 of the following respiratory signs/symptoms: cough, shortness of breath or difficulty breathing, or clinical or radiographical evidence of pneumonia; and had at least 1 nasopharyngeal swab, nasal swab, or saliva sample (or respiratory sample, if hospitalized) positive for SARS-CoV-2.
Time Frame: Day 43 (14 days after second injection) up to 2.5 months after second injection
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: mRNA-1273 100 μg | Part 1A: Placebo
Number analyzed (Participants) | 2142 | 1044
Participants | 0 | 6
Statistical Analysis 1: Comparison: Part 1A: mRNA-1273 100 μg vs Part 1A: Placebo; Test type: Other; VE; VE (percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo); VE = 100.0, 95% CI 2-sided [lower limit 61.2] (NA = not estimable (not reached).) — The 95% CI of the ratio was calculated using the exact method conditional upon the total number of cases, adjusting for person-years

16. Secondary Outcome: Part 1A Number of Participants With Secondary Case Definition of COVID-19 (Center for Disease Control and Prevention [CDC] Case Definition)
Description: Secondary case definition of COVID-19 was defined by the following criteria: 1 systemic or respiratory symptoms: fever (temperature > 38ºC/≥ 100.4ºF), or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle aches, or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea, or vomiting or diarrhea, and at least one positive test for SARS-CoV-2.
Time Frame: Day 43 (14 days after second injection) up to a median follow up of 2.5 months after second injection
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: mRNA-1273 100 μg | Part 1A: Placebo
Number analyzed (Participants) | 2142 | 1044
Participants | 2 | 9
Statistical Analysis 1: Comparison: Part 1A: mRNA-1273 100 μg vs Part 1A: Placebo; Test type: Other — [test comment as in outcome 13, analysis 1]; VE; VE (percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo); VE = 89.9, 95% CI 2-sided [51.0 to 98.9]

17. Secondary Outcome: Part 1C-1 SRR of the Post-booster Serum Binding Antibody (bAb) Against Variants of Interest (B.1.1.7, B.1.351, B.1.617.2, and P.1) as Measured by MSD
Description: Percentage of participants with seroresponse for bAb measured using (MesoScale Discovery) MSD are reported. Seroresponse from baseline (pre-Dose 1) at a participant level was defined as a change from below the LLOQ to equal or above 4 * LLOQ, or at least a 4-fold-rise if baseline (pre-Dose 1) is equal to or above the LLOQ.
Time Frame: BD Day 29
Population: Part 1C-1 PPIS: participants were baseline (pre-dose 1 of Part 1A) SARS-CoV-2 negative, had BD-Day 1 and BD-Day 29 Ab assessment, had no major protocol deviations, did not receive off-study COVID-19 vaccination prior to BD-Day 29 visit, received 2 doses of mRNA-1273 in the Blinded Phase per schedule, and received BD. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1C-1: mRNA-1273 50 µg BD
Number analyzed (Participants) | 324
Percentage of participants
  B.1.1.7 | 100.0 (98.9) [98.9 to 100.0]
  B.1.351 | 100.0 (98.9) [98.9 to 100.0]
  B.1.617.2 | 100.0 (98.9) [98.9 to 100.0]
  P.1 | 100.0 (98.9) [98.9 to 100.0]

18. Secondary Outcome: Part 1C-1 GMC of Post-booster Pseudovirus nAb Against Variant Strain (B.1.1.529)
Description: Post-booster Pseudovirus nAb against B.1.1.529 (LLOQ: 8 AU/mL, ULOQ: 24503 AU/mL). Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available.
Time Frame: BD Day 29
Population: Part 1C-1 PPIS: participants were baseline (pre-dose 1 of Part 1A) SARS-CoV-2 negative, had BD-Day 1 and BD-Day 29 Ab assessment, had no major protocol deviations, did not receive off-study COVID-19 vaccination prior to BD-Day 29 visit, received 2 doses of mRNA-1273 in the Blinded Phase per schedule, and received BD. Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1C-1: mRNA-1273 50 µg BD
Number analyzed (Participants) | 331
AU/mL | 943.4 (853.5) [853.5 to 1042.8]

19. Secondary Outcome: Part 3 SRR of Serum Pseudovirus nAb Post Dose 1 of mRNA-1273.222 Against Omicron BA.4/BA.5 Compared With Those From Young Adult (18 to 25 Years of Age) Vaccine Recipients (Day 57) in Study P301
Description: Seroresponse from pre Dose 1 Baseline at a participant level was defined as a change from below the LLOQ to equal or above 4 * LLOQ, or at least a 4-fold rise if Baseline was equal to or above the LLOQ (LLOQ: 103 AU/mL, ULOQ:
  28571 AU/mL). PPIS P301: randomly selected participants from Study P301 aged 18-25 meeting pre-specified criteria and SARS-CoV-2 negative were used for comparison of immune response.
Time Frame: Day 29 Study P203/Day 57 Study P301
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3: mRNA-1273.222 50 µg | Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg
Number analyzed (Participants) | 372 | 294
percentage of participants | 95.4 [92.8 to 97.3] | 0.0 [0.0 to 1.2]

20. Secondary Outcome: Part 3 Pseudovirus nAb SRR of Post Dose 1 of mRNA-1273.222 Against Ancestral Strain Compared With Those From Young Adult (18 to 25 Years of Age) Vaccine Recipients (Day 57) in Study P301
Description: Percentage of participants with seroresponse for pseudovirus nAb measured using PsVNA assay are reported. Seroresponse from pre Dose 1 Baseline at a participant level was defined as a change from below the LLOQ to equal or above 4 * LLOQ, or at least a 4-fold rise if Baseline was equal to or above the LLOQ. PPIS P301: randomly selected participants from Study P301 aged 18-25 meeting pre-specified criteria and SARS-CoV-2 negative were used for comparison assessments of immune response.
Time Frame: Day 29 P203/Day 57 P301
Population: Part 3 PPIS-Pos: participants who received Dose 1 of mRNA-1273.222, had Day 29 antibody assessments, no major protocol deviations, did not receive off-study COVID-19 vaccination prior to Day 29, and were SARS-CoV-2 positive at baseline. 'Overall number of participants analyzed' = participants evaluable for the endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3: mRNA-1273.222 50 µg | Study mRNA-1273-P301 (NCT04470427 ) mRNA-1273 100 μg
Number analyzed (Participants) | 370 | 295
percentage of participants | 94.9 [92.1 to 96.9] | 99.3 [97.6 to 99.9]

21. Secondary Outcome: Part 3 GM Value of Post Dose 1 (Day 29) of mRNA-1273.222 bAb Against Other Variants of Interest
Description: mRNA-1273.222 bAb was measured using a S-binding IgG immunoassay. Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ are replaced by the ULOQ if actual values are not available (LLOQ: 397 AU/ml, ULOQ: 2200000 AU/mL).
Time Frame: Day 29
Population: Part 3 PPIS: all participants who received Dose 1 of mRNA-1273.222 and had both Baseline (pre Dose 1) and Day 29 antibody assessment, had no major protocol deviations that impacted key or critical data; and had not received off-study COVID-19 vaccination prior to Day 29. 'Overall number of participants analyzed' = participants evaluable for the endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 3: mRNA-1273.222 50 µg
Number analyzed (Participants) | 372
AU/mL
  BA.5 | 282734.2 [266581.0 to 299866.1]
  AY.4 | 557963.4 [529270.6 to 588211.6]
  B.1.1.7 | 434879.0 [412699.2 to 458250.8]
  B.1.351 | 431476.5 [409656.1 to 454459.1]
  B.1.1.529 | 189826.0 [178578.0 to 201782.5]
  P.1 | 471868.9 [446431.3 to 498756.0]

22. Secondary Outcome: Part 1C-2 GM Value of mRNA-1273 Booster Against Variants of Interest at Day 29
Time Frame: Day 29
Population: As a result of emergence of a more divergent variant of concern (Omicron), Part 1C-2 enrollment and booster dosing were discontinued. Therefore, data were collected for Part 1C-2 Primary Outcome Measure but after Part 1C-2 was discontinued, per Sponsor, it was decided that data would not be collected for this Part 1C-2 Secondary Outcome Measure and instead collect data for the more updated variant containing vaccine (Part 3: mRNA-1273.222).
Arm/Group | Part 1C-2: mRNA-1273 50 μg BD
Number analyzed (Participants) | 0

23. Secondary Outcome: Part 1A GM Level of SARS-CoV-2 Spike Protein-specific bAb at Days 1, 57, 209, 394
Description: SARS-CoV-2 Spike Protein-specific bAb were measured using MSD electrochemiluminescence multiplex assay. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ are replaced by the ULOQ if actual values are not available (LLOQ: 69 AU/mL, ULOQ: 14400000 AU/mL).
Time Frame: Days 1, 57, 209, 394
Population: Part 1A PPIS for long term analysis included all randomized participants who had a negative SARS-CoV-2 status at baseline (pre-Dose 1), received planned doses of study drug per schedule, complied with immunogenicity testing schedule, and had no major protocol deviations that impacted key or critical data. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1A: mRNA-1273 100 μg
Number analyzed (Participants) | 369
AU/mL
  Day 1 | 65.848 [60.348 to 71.850]
  Day 57: number analyzed (Participants) | 366
  Day 57 | 346830.736 [330758.387 to 363684.079]
  Day 209: number analyzed (Participants) | 366
  Day 209 | 79624.290 [73959.321 to 85723.172]
  Day 394: number analyzed (Participants) | 356
  Day 394 | 58647.246 [52309.921 to 65752.336]

24. Secondary Outcome: Part 1A GM Value of SARS-CoV-2-Specific nAb at Days 1, 57, 209, 394
Description: SARS-CoV-2-Specific nAb were measured using PsVNA assay. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ are replaced by the ULOQ if actual values are not available (LLOQ: 10 AU/mL, ULOQ: 281600 AU/mL).
Time Frame: Days 1, 57, 209, 394
Population: Part 1A PPIS for long term analysis included all randomized participants who had a negative SARS-CoV-2 status at baseline (pre-Dose 1), received planned doses of study drug per schedule, complied with immunogenicity testing schedule, and had no major protocol deviations that impacted key or critical data. 'Overall number of participants analyzed' = participants evaluable for this endpoint. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1A: mRNA-1273 100 μg
Number analyzed (Participants) | 369
AU/mL
  Day 1 | 11.249 [10.712 to 11.812]
  Day 57: number analyzed (Participants) | 366
  Day 57 | 1868.363 [1758.809 to 1984.742]
  Day 209: number analyzed (Participants) | 366
  Day 209 | 625.363 [583.319 to 670.437]
  Day 394: number analyzed (Participants) | 363
  Day 394 | 550.262 [489.875 to 618.093]

25. Secondary Outcome: Part 1C-1 GM Value of Post-booster Dose Serum bAb Against Variants of Interest (B.1.1.7, B.1.351, B.1.617.2, and P.1) as Measured by MSD
Description: Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. B.1.1.7 (LLOQ: 52, ULOQ: 8800000), B.1.351 (LLOQ: 111, ULOQ: 5000000), B.1.617.2 (LLOQ: 49, ULOQ: 7400000), P.1 (LLOQ: 143, ULOQ: 5800000).
Time Frame: BD Day 29
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1C-1: mRNA-1273 50 µg BD
Number analyzed (Participants) | 324
AU/mL
  B.1.1.7 | 581097.8 (543987.7) [543987.7 to 620739.5]
  B.1.351 | 431569.2 (404983.2) [404983.2 to 459900.6]
  B.1.617.2 | 456423.3 (429083.9) [429083.9 to 485504.8]
  P.1 | 417277.2 (391682.5) [391682.5 to 444544.5]

26. Other Pre Specified Outcome: Number of Deaths Related to Study Drug
Description: A death that occurred during the study or that came to the attention of the investigator during the study was reported to the Sponsor, whether or not it was considered related to study drug. The investigator assessed causality (that is, whether there is a reasonable possibility that the study drug caused the death). The relationship was characterized using the following classifications: Not related: There was not a reasonable possibility of a relationship to the study drug. The temporal sequence of the death relative to administration of the study drug was not reasonable and/or the death was more likely explained by a cause other than the study drug. Related: There was a reasonable possibility of a relationship to the study drug. There was evidence of exposure to the study drug. The temporal sequence of the death relative to the administration of the study drug was reasonable. The death was more likely explained by the study drug than by another cause.
Time Frame: Day 1 up to Day 751
Population: Safety Set: participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1B: mRNA-1273 100 µg: Participants previously received 2 doses of placebo in the blinded phase and then received crossover vaccination with 100 μg of mRNA-1273.
- Part 3: mRNA-1273.222 50 ug Second Dose: Participants received 1 dose of mRNA-1273.222 50 µg by IM injection (Day 1) and a second dose approximately 6 months after the first dose (Day 181).
Arm/Group | Part 1A: mRNA-1273 100 μg | Part 1A: Placebo | Part 1B: mRNA-1273 100 µg | Part 1C-1: mRNA-1273 50 µg BD | Part 1C-2: mRNA-1273 50 μg BD | Part 2: mRNA-1273 50 μg | Part 2: mRNA-1273 50 μg BD | Part 3: mRNA-1273.222 50 μg 1 Dose | Part 3: mRNA-1273.222 50 ug Second Dose
Number analyzed (Participants) | 2486 | 1240 | 96 | 1408 | 155 | 52 | 19 | 388 | 335
Participants
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Deaths related to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 751
Description: All-cause mortality: enrolled; AEs: participants received at least 1 dose of study drug.
  Non-serious SARs persisting beyond 7 days, leading to discontinuation, or medically attended were classified as unsolicited AEs in Part 1/2 but not in Part 3. COVID-19/SARS-CoV-2 infections were AEs in Part 1/2 but were considered clinical events for efficacy in Part 3 and not AEs.
Groups:
- Part 1A: Placebo: Participants received at least 1 of 2 doses of placebo by IM injection (Day 1 and Day 29).
- Part 2: mRNA-1273 50 ug BD: Participants received open-label mRNA-1273 50 µg in Part 2 and then a single BD of 50 μg mRNA-1273 IM injection on BD Day 1 in Part 2.
- Part 3: mRNA1273.222 50 µg 1 Dose: Participants received 1 dose of mRNA-1273.222 50 µg by IM injection (Day 1).
Arm/Group | Part 1A: mRNA-1273 100 μg | Part 1A: Placebo | Part 1B: mRNA-1273 100 µg | Part 1C-1: mRNA-1273 50 µg BD | Part 1C-2: mRNA-1273 50 μg BD | Part 2: mRNA-1273 50 μg | Part 2: mRNA-1273 50 ug BD | Part 3: mRNA1273.222 50 µg 1 Dose | Part 3: mRNA-1273.222 50 ug Second Dose
All-Cause Mortality (participants affected / at risk) | 0/2486 | 0/1240 | 0/96 | 0/1408 | 0/155 | 0/52 | 0/19 | 0/388 | 1/335
Serious Adverse Events (participants affected / at risk) | 21/2486 | 4/1240 | 2/96 | 9/1408 | 3/155 | 0/52 | 0/19 | 12/388 | 4/335
Other Adverse Events (participants affected / at risk) | 943/2486 | 155/1240 | 22/96 | 429/1408 | 28/155 | 12/52 | 7/19 | 77/388 | 51/335
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A: mRNA-1273 100 μg (N=2486) | Part 1A: Placebo (N=1240) | Part 1B: mRNA-1273 100 µg (N=96) | Part 1C-1: mRNA-1273 50 µg BD (N=1408) | Part 1C-2: mRNA-1273 50 μg BD (N=155) | Part 2: mRNA-1273 50 μg (N=52) | Part 2: mRNA-1273 50 ug BD (N=19) | Part 3: mRNA1273.222 50 µg 1 Dose (N=388) | Part 3: mRNA-1273.222 50 ug Second Dose (N=335)
Pectus excavatum (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syringomyelia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Investigator and Sponsor assessment of drug-induced liver injury was not related to study drug.
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Investigator and Sponsor assessment of anaphylactic reaction was not related to study drug due to long time to onset (171 days).
Amoebic dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Murine typhus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — AE of gunshot wound resulted in death. Investigator assessment was not related to study drug.
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Status migrainosus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Idiopathic generalised epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Obstructive nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Sponsor assessment of AE of hypercoagulation was not related to study drug based on medical history, results of the heart biopsy, including findings of long-standing pre-existing heart failure and long time to onset (256 days).
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Sponsor assessment of AE of cardiogenic shock was not related to study drug based on medical history, results of the heart biopsy, including findings of long-standing pre-existing heart failure and long time to onset (256 days).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A: mRNA-1273 100 μg (N=2486) | Part 1A: Placebo (N=1240) | Part 1B: mRNA-1273 100 µg (N=96) | Part 1C-1: mRNA-1273 50 µg BD (N=1408) | Part 1C-2: mRNA-1273 50 μg BD (N=155) | Part 2: mRNA-1273 50 μg (N=52) | Part 2: mRNA-1273 50 ug BD (N=19) | Part 3: mRNA1273.222 50 µg 1 Dose (N=388) | Part 3: mRNA-1273.222 50 ug Second Dose (N=335)
Abdominal pain (Gastrointestinal disorders) | 8 (9) | 3 (3) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injection site lymphadenopathy (General disorders) | 137 (146) | 6 (6) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 11 (12) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 26 (34) | 22 (30)
Parainfluenzae virus infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 60 (64) | 6 (6) | 4 (4) | 16 (17) | 0 (0) | 0 (0) | 0 (0) | 30 (34) | 23 (26)
Influenza (Infections and infestations) | 19 (20) | 0 (0) | 1 (1) | 30 (30) | 7 (8) | 1 (1) | 2 (2) | 5 (6) | 0 (0)
COVID-19 (Infections and infestations) | 382 (383) | 34 (35) | 11 (11) | 257 (267) | 10 (10) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 81 (82) | 25 (25) | 6 (6) | 39 (39) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 41 (41) | 6 (6) | 0 (0) | 14 (14) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 58 (60) | 3 (3) | 1 (1) | 26 (27) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 117 (129) | 51 (57) | 1 (1) | 28 (29) | 1 (1) | 1 (1) | 0 (0) | 20 (27) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 257 (293) | 28 (32) | 3 (3) | 81 (101) | 6 (8) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Tooth abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Part 1C-2 enrollment discontinued before planned number of participants. Part 2 discontinued early due to availability of updated variant vaccine (mRNA-1273.222); no hypothesis testing done for primary endpoint/other endpoints not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT04649151/Prot_001.pdf
  • Statistical Analysis Plan (2024-06-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT04649151/SAP_002.pdf
  • Informed Consent Form (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT04649151/ICF_003.pdf